CLINICAL TRIAL: NCT00753974
Title: Cardiovascular Biorepository
Status: Enrolling by invitation | Type: Observational
Sponsor: Kenneth S. Campbell (Other)
Responsible Party: Sponsor-Investigator, Kenneth S. Campbell, PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 46103
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens procured include myocardium from left and right atria, left and right ventricle, and septum, aortic wall, and venous blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- biological specimen: Biological specimen is taken from cardiovascular procedures that would have been discarded

SUMMARY:
Use biospecimens procured from patients and organ donors to improve understanding of molecular, cellular, and tissue-level processes produced by cardiovascular disease and therapeutic interventions

DETAILED DESCRIPTION:
This is a prospective evaluation of patients undergoing cardiovascular procedures at the University of Kentucky Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiovascular surgery/procedure at the University of Kentucky who are at least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • All patients undergoing cardiovascular surgery/procedure at the University of Kentucky who are at least 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-06; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Use biospecimens procured from patients and organ donors to improve understanding of molecular, cellular, and tissue-level processes produced by cardiovascular disease and therapeutic interventions. | 6/26/2008 - 6/9/2030
  This research aims to advance understanding of cardiovascular disease and to support the development of improved therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Campbell, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Department of Internal Medicine, Division of Cardiovascular Medicine, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No